CLINICAL TRIAL: NCT04003870
Title: Controlled Trial to Compare the Achilles Tendon Load During Running in Flatfeet Subjects Using a Customized Arch Support Orthoses vs an Orthotic Heel Lift
Brief Title: Orthotics and Achilles Load in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North District Hospital (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor of Orthopaedics and Traumatology, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUHK
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Achilles Tendinopathy; Flatfoot; Sports Injury
MeSH Terms: conditions — Flatfoot; Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Runner (Experimental): Subject will undergo an assessment wearingeither the CASO or the HL. Sequence of CASO of HL will be randomly allocated.
  Interventions: Device: CASO; Device: HL

INTERVENTIONS:
Device: CASO — Customized arch support orthoses (CASO)
Device: HL — Orthotic Heel Lift (HL)

SUMMARY:
Compare Customized arch support orthoses (CASO) and orthotic heel lift (HL) on the effect of ATL in recreational runners with pronated feet.

DETAILED DESCRIPTION:
This was a controlled laboratorial, within subject, repeated measures study. The aim of this study was to compare two clinically applied treatment options: Customized arch support orthoses (CASO) and orthotic heel lift (HL) on the effect of ATL in recreational runners with pronated feet. It implicated to provide a better understanding of the types of foot orthoses for flatfeet runners and additional biomechanical evidence for the clinical field to guide orthotic prescription as well as selection for Achilles tendinopathy management.

ELIGIBILITY:
Inclusion:

* Foot Posture Index (FPI) was used as evaluating pronated foot posture. Subjects with FPI scores of 6-12 were recruited in the current study.
* All participants should be free of Achilles tendinopathy and triceps surae injury for 6 months.
* no previous surgery.
* not previously attempted any foot orthoses intervention before this study.

Exclusion:

* leg-length discrepancy
* rigid forefoot varus deformity
* gastrocnemius equinus
* structural hallux limitus, or rigidus
* Any musculoskeletal or neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Peak plantarflexion moment | Day 0
  8-camera motion capturing system
Peak Achilles tendon load | Day 0
  Piezoelectric force platform, computed using the Newton-Euler inverse-dynamics

CONTACTS AND LOCATIONS:
Locations (1):
- CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee KKW, Ling SKK, Yung PSH. Controlled trial to compare the Achilles tendon load during running in flatfeet participants using a customized arch support orthoses vs an orthotic heel lift. BMC Musculoskelet Disord. 2019 Nov 13;20(1):535. doi: 10.1186/s12891-019-2898-0. PMID 31722697
- See also: Related Info — https://rdcu.be/b38yd